CLINICAL TRIAL: NCT04568122
Title: Rapid Turnaround, Home-based Saliva Testing for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: BioBox (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 58629
Record Dates: First submitted 2020-09-25; First posted 2020-09-29 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Enrollment is to a single group. Specific eligibility criteria apply depending on whether the participant is a hospitalized patient, in high-risk or infected population, or low-risk population
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Saliva test (Experimental): Participants perform each test assay, noting the results for comparison by technician, and completing survey questionnaires.
  Interventions: Device: Saliva test kit

INTERVENTIONS:
Device: Saliva test kit — Kit including tube with closed reagents using loop-mediated isothermal amplification (LAMP) assay to detect SARS-CoV-2 virus.
  Other Names: SnapDx

SUMMARY:
The aim of the study is to demonstrate the feasibility and validity of a saliva based home surveillance monitoring test for SARS-CoV-2 infection.

Participants will be asked to carry out as many tests as are included in the bag they are provided, on a daily basis until they are used up.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients

  * Hospitalized at Stanford Health Care for COVID-related complications and tested positive for SARS-CoV-2 with a PCR-based test
  * Able to understand and consent to study and with a clinical trajectory likely to be consistent with multi-day participation
* High-risk/positive population

  * Seeking testing for suspected COVID or a participant in a study of COVID-positive outpatients
  * Own an internet-enabled phone or device capable of loading web pages, receiving text messages, and taking/uploading photos.
  * Willing to participate in the study for 6 months
* Low-risk population

  * Own an internet-enabled phone or device capable of loading web pages, receiving text messages, and taking/uploading photos.
  * Willing to participate in the study for 6 months

Exclusion Criteria:

* All participants:

  * Participants with salivary gland dysfunction (including patients with Sjogren's disease or those with xerostomia associated with lupus or rheumatoid arthritis)
  * Participants will not be eligible if they identify any reason they are unable to participate in the study
* High-risk/positive population

  * Participants who have color blindness
  * Participants unable to operate the SnapDx device
* Low-risk population

  * Participants with prior confirmed SARS-CoV-2 infection
  * Participants who have color blindness
  * Participants unable to operate the SnapDx device

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1277 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manu Prakash, PhD, Principal Investigator — Stanford University; Manisha Desai, PhD, Principal Investigator — Stanford University; Euan A Ashley, MRCP, DPhil, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - SHC Valley Care, Pleasanton, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: https://www.snapdx.org/ (for more information and how to enroll) — https://www.snapdx.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1277 participants signed consent; 353 were allocated to a study arm: participants who came to the study site to collect a kit (First, Second, and Third Distribution groups) or provided saliva samples (Positive Saliva Collection and Negative Saliva Collection groups).
Groups:
- Saliva Test - First Distribution; Saliva Test - Second Distribution: Participants provide two test samples at home using the saliva test kit to detect the SARS-CoV-2 virus.
- Saliva Test - Third Distribution: Participants provide one test sample at study visit using the saliva test kit to detect the SARS-CoV-2 virus.
- Positive Saliva Collection: Participants provide one saliva sample confirmed positive for SARS-CoV-2 virus used in lab to validate device function.
- Negative Saliva Collection: Participants provide one saliva sample confirmed negative for SARS-CoV-2 virus used in lab to validate device function.
Period: Overall Study
Arm/Group | Saliva Test - First Distribution | Saliva Test - Second Distribution | Saliva Test - Third Distribution | Positive Saliva Collection | Negative Saliva Collection
Started | 94 | 112 | 135 | 9 | 3
Completed One Test | 46 | 68 | 131 | 9 | 3
Completed 2 Tests | 32 | 53 | 0 | 0 | 0
Completed | 46 | 68 | 131 | 9 | 3
Not Completed | 48 | 44 | 4 | 0 | 0
Not completed — Lost to Follow-up | 48 | 44 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saliva Test - First Distribution | Saliva Test - Second Distribution | Saliva Test - Third Distribution | Positive Saliva Collection | Negative Saliva Collection | Total
Number analyzed (Participants) | 94 | 112 | 135 | 9 | 3 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (15.8) | 46.8 (20.6) | 52.6 (17.0) | 23.8 (5.1) | 24.3 (5.51) | 46.11 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 73 | 91 | 8 | 3 | 217
  Male | 52 | 39 | 44 | 1 | 0 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 20 | 10 | 0 | 0 | 53
  Not Hispanic or Latino | 66 | 91 | 124 | 9 | 3 | 293
  Unknown or Not Reported | 5 | 1 | 1 | 0 | 0 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race category options in patient-completed online survey
  Participants
    Asian | 13 | 24 | 21 | 4 | 2 | 64
    Black or African American | 3 | 2 | 1 | 0 | 0 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 5 | 0 | 0 | 0 | 5
    White | 60 | 65 | 103 | 5 | 1 | 234
    More than one race | 6 | 8 | 0 | 0 | 0 | 14
    Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 2
    Other | 10 | 8 | 10 | 0 | 0 | 28
Region of Enrollment [Number; unit: participants]
  United States | 94 | 112 | 135 | 9 | 3 | 353

OUTCOME MEASURES:

1. Primary Outcome: Number of Matched Test Colormetric Interpretation as a Measure of Interrater Reliability
Description: Feasibility Outcome. Discrepancy in interpretation of colormetric readout by participant versus by technician via photo. Passed test = void of manufacturing or user error.
Time Frame: Up to 5 days per participant
Population: Data were collected from the Saliva Test - First, Second, and Third Distribution groups only. Participants who completed at least one test are included in the analysis.
Measure: Count of Units; unit: Completed tests
Units Other Than Participants: Completed tests
Arm/Group | Saliva Test - First Distribution | Saliva Test - Second Distribution | Saliva Test - Third Distribution
Number analyzed (Participants) | 46 | 68 | 131
Number analyzed (Completed tests) | 78 | 121 | 131
Completed tests
  Total passed tests | 52 | 69 | 97
  Matching interpretation | 27 | 67 | 93

2. Primary Outcome: Number of Positive Home Saliva Tests as Determined by the Patient
Description: Validity Outcome.
Time Frame: Up to 5 days per participant
Population: as for outcome 1
Measure: Count of Units; unit: Completed tests
Units Other Than Participants: Completed tests
Arm/Group | Saliva Test - First Distribution | Saliva Test - Second Distribution | Saliva Test - Third Distribution
Number analyzed (Participants) | 46 | 68 | 131
Number analyzed (Completed tests) | 78 | 121 | 131
Completed tests | NA — Data were not analyzable for this outcome because reagents were not stable over the course of a day and the dye used was too sensitive to pH, leading to unreliable data. | NA — Data were not analyzable for this outcome because reagents were not stable over the course of a day and the dye used was too sensitive to pH, leading to unreliable data. | NA — Data were not analyzable for this outcome because reagents were not stable over the course of a day and the dye used was too sensitive to pH, leading to unreliable data.

3. Secondary Outcome: Participant-rated Confidence in Interpreting Results
Description: Validity Outcome (ease of interpretation). Number of participants responding by category when asked to provide a rating on being "Confident in Interpreting Results."
Time Frame: Up to 5 days per participant
Population: Data were collected for the Third Distribution group only; participants who completed the test are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Saliva Test - Third Distribution
Number analyzed (Participants) | 131
Participants
  Strongly agree | 53
  Agree | 61
  Somewhat agree | 9
  Neither agree nor disagree | 2
  Somewhat disagree | 3
  Disagree | 3
  Strongly disagree | 0

4. Secondary Outcome: Participant-rated Ease of Use
Description: Validity Outcome (ease of use). Number of participants responding by category when asked to provide a rating on SnapDx being "Easy to Learn to Use."
Time Frame: Up to 5 days per participant
Population: Data were collected for the First, Second, and Third distribution groups only; participants who completed the test and responded to the survey question are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Saliva Test - First Distribution | Saliva Test - Second Distribution | Saliva Test - Third Distribution
Number analyzed (Participants) | 29 | 64 | 131
Participants
  Strongly agree | 0 | 5 | 13
  Agree | 6 | 22 | 52
  Somewhat agree | 7 | 10 | 39
  Neither agree nor disagree | 2 | 4 | 4
  Somewhat disagree | 8 | 12 | 18
  Disagree | 3 | 6 | 5
  Strongly disagree | 3 | 5 | 0

5. Secondary Outcome: Number of Participants That Called Technical Support
Description: Feasibility Outcome (ease of use). Number of participants that called technical support, by reason (e.g., processing was not possible due to broken part).
Time Frame: Up to 5 days per participant
Population: Data were collected for this outcome from the Saliva Test - First and Second distribution groups only.
Measure: Count of Participants; unit: Participants
Arm/Group | Saliva Test - First Distribution | Saliva Test - Second Distribution
Number analyzed (Participants) | 94 | 112
Participants | 0 | 0

6. Secondary Outcome: Sample Integrity
Description: Feasibility Outcome. The participants were asked to determine whether the saliva sample filled up to the indicated line, and if there were bubbles present as a measure of sample integrity.
Time Frame: Up to 5 days per participant
Population: Data were collected from the Saliva Test - First and Third distribution groups only. Participants who completed at least one test are included in the analysis.
Measure: Count of Units; unit: Test samples
Units Other Than Participants: Test samples
Arm/Group | Saliva Test - First Distribution | Saliva Test - Third Distribution
Number analyzed (Participants) | 46 | 131
Number analyzed (Test samples) | 78 | 131
Test samples
  Sufficient sample | 78 | 131
  Significant presence of bubbles | 25 | 50

7. Secondary Outcome: Sensitivity of Sample Test Kit
Description: Validity Outcome. Analysis of saliva samples provided by participants and run through sample test kit by study lab. Sensitivity = number of true positives out of the positive tests run. Samples may have been split and run through more than one test.
Time Frame: Up to 5 days per participant
Population: Data were collected from the Validation Saliva Samples group only.
Measure: Count of Units; unit: Positive tests run
Units Other Than Participants: Positive tests run
Arm/Group | Positive Saliva Collection
Number analyzed (Participants) | 9
Number analyzed (Positive tests run) | 5
Positive tests run | 4

8. Secondary Outcome: Specificity of Sample Test Kit
Description: Validity Outcome. Analysis of saliva samples provided by participants and run through sample test kit by study lab. Specificity = number of true negatives out of negative tests run. Samples may have been split and run through more than one test.
Time Frame: Up to 5 days per participant
Population: Specificity analysis includes samples confirmed negative from the First or Second Distribution groups, and samples from the Negative Saliva Collection group only
Measure: Count of Units; unit: Negative tests run
Units Other Than Participants: Negative tests run
Groups:
- Negative Sample Analysis: Confirmed negative samples collected from participants in the First and Second Distribution groups used for specificity analysis.
- All Samples: All positive saliva samples.
Arm/Group | Negative Sample Analysis | Negative Saliva Collection | All Samples
Number analyzed (Participants) | 206 | 3 | 209
Number analyzed (Negative tests run) | 18 | 10 | 28
Negative tests run | 15 | 10 | 25

ADVERSE EVENTS:
Time Frame: Average approximately 1 week
Arm/Group | Saliva Test - First Distribution | Saliva Test - Second Distribution | Saliva Test - Third Distribution | Positive Saliva Collection | Negative Saliva Collection
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/112 | 0/135 | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/112 | 0/135 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 0/94 | 0/112 | 0/135 | 0/9 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT04568122/Prot_SAP_000.pdf